CLINICAL TRIAL: NCT05639790
Title: The Effectiveness of Using E-Cigarettes as Harm Reduction Strategy for Smoking Cessation and Decreasing Risk of Diseases Among Heavy Smokers: an Open-label Randomized Controlled Trial
Brief Title: The Effectiveness of Using E-Cigarettes for Smoking Cessation and Decreasing Risk of Diseases Among Heavy Smokers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to issues arised from the collaboration contract between sponsor and research site
Sponsor: Shenzhen Smoore Technology Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SR20221001
Record Dates: First submitted 2022-11-03; First posted 2022-12-06 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counselling (Sham Comparator): Health counselling from a licensed mental health counselor
  Interventions: Other: Health Counselling
- Eletronic cigarette (Experimental): Ad libitum use of electronic cigarettes for 1 month and health counselling from a licensed mental health counselor
  Interventions: Combination Product: Electronic cigarettes + Health Counselling; Other: Health Counselling

INTERVENTIONS:
Combination Product: Electronic cigarettes + Health Counselling — Ad libitum use of electronic cigarettes for 1 month
  Arms: Eletronic cigarette
Other: Health Counselling — Health Counselling from a licensed mental health counselor

SUMMARY:
The goal of this clinical trial is to evaluate effectiveness of using e-cigarettes as harm reduction strategy for smoking cessation and decreasing risk of diseases in heavy smokers. The main questions it aims to answer are:

* Is there any effectiveness of using E-cigarette as a harm reduction strategy for smoking cessation?
* what are the impacts of using E-cigarette on respiratory function and risk of COPD?
* Assess the exposure to harmful and potential harmful constituents (HPHCs) of using E-cigarette

Participants will be randomized into a 6 months single-center, open label trial comparing study outcomes among 2 arms: health counselling, E-cigarette + health counselling. The EC arm will receive EC for 1 month. All 2 arms will receive health counselling from a licensed mental health counselor. After baseline, participants will report their use of combustible cigarette in both arms and EC use in the EC arm every day via online questionnaire in Wechat for behavioral monitoring.

If there is a comparison group: Researchers will compare health counselling group to see if E-cigarrette intervention is an effective way to stop smoking, and if there any change in respiratory function and change in exposure to harmful and potential harmful constituents (HPHCs).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years old, gender is not limited
* The nicotine dependence test (FNDT) result score is 6-10 points
* Self-reported smoking at least 10 cigarettes a day, and smoking for at least 3 years
* Self-reported no current willingness to quit smoking
* Self-reported difficulty controlling the need to smoke, or smoking while sick in bed
* Must not accepted smoking cessation treatment in the last 3 months according to the self-report
* Must have never tried e-cigarette before
* Must be able to fully understand the purpose, nature and content of the research, and voluntarily sign the informed consent form as a subject
* Must agree and able to communicate well with the researcher, and able to complete the online questionnaire and examination in accordance with the research regulations.

Exclusion Criteria:

* Self-reported pregnant or breastfeeding
* Severe disease (defined as an illness or condition that put the patient at risk, interfere the trial results, or affect the patient's ability to participate in the trial judged by the panel)
* Past diagnosis of COPD, lung cancer, pneumoconiosis, bronchiectasis, interstitial lung disease, bronchial asthma, or other restrictive ventilatory disorder
* Living with severe heart, brain, liver, kidney, blood system diseases or malignant tumors
* Moderate-severe renal impairment, or creatinine clearance (CCr) ≤50ml/min
* Phenylpyruvaturia
* Allergic predisposition (be allergic to two or more substances), and is allergic to any of the components in e-cigarettes or e-liquid (e.g., benzoic acid, propylene glycol, glycerin, nicotine, etc.)
* Already been enrolled into a smoking cessation treatment, including but not limited to nicotine replacement therapy (NRT), varenicline, bupropion
* Living with mental illness, a history of chronic alcoholism, drug abuse, or any factor that affects compliance
* Participating in other clinical trials
* Life-threatening condition with a life expectancy less than 1 year
* Researcher believes that it is not suitable to participate in this researcher.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence abstinence | 1 month
  The effectiveness of smoking cessation with intervention

SECONDARY OUTCOMES:
Score of COPD-SQ questionnaire | 1 month
  self-reported score of COPD-SQ questionnaire
Score of COPD-PS questionnaire | 1 month
  self-reported score of COPD-PS questionnaire
Score of mMRC scale | 1 month
  self-reported score of modified Medical Research Council scale
Score of CAT questionnaire | 1 month
  self-reported score of COPD Assessment Test
%ratio of FEV1/FVC | 1 month
  the proportion of a person's vital capacity that are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC).
Concentration of 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) | 1 month
  Concentration of 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) in urine
Concentration of 3-Hydroxypropyl- mercapturic acid (3-HPMA) | 1 month
  Concentration of 3-Hydroxypropyl- mercapturic acid (3-HPMA) in urine
Concentration of 2-Cyanoethylmercaturic acid (CEMA) | 1 month
  Concentration of 2-Cyanoethylmercaturic acid (CEMA) in urine
Concentration of S-phenylmercapturic Acid (S-PMA) | 1 month
  Concentration of S-phenylmercapturic Acid (S-PMA) in urine
Concentration of 3-Hydroxy-1-methylpropyl-mercapturic acid (3-HMPMA) | 1 month
  Concentration of 3-Hydroxy-1-methylpropyl-mercapturic acid (3-HMPMA) in urine
Concentration of N-nitrosonornicotine (NNN) | 1 month
  Concentration of N-nitrosonornicotine (NNN) in urine
Concentration of S-benzyl-mercapturic acid (S-BMA) | 1 month
  Concentration of S-benzyl-mercapturic acid (S-BMA) in urine
Concentration of cotinine | 1 month
  Concentration of cotinine in urine
Concentration of Trans-3-Hydroxy Cotinine (TNE-2) | 1 month
  Concentration of Trans-3-Hydroxy Cotinine (TNE-2) in urine
Concentration of total Nicotine equivalent | 1 month
  Concentration of total Nicotine equivalent in urine
Concentration of formic acid | 1 month
  Concentration of formic acid in urine

IPD SHARING:
Plan to Share IPD: No